CLINICAL TRIAL: NCT06592456
Title: Immunogenicity and Safety of a Live Attenuated Varicella Vaccine in Adolescents and Adults Aged Between 13 to 55 Years : a Double-Blind, Randomized, Parallel-Controlled Phase III Clinical Trial in China
Brief Title: A Phase III Clinical Trial Assessing the Immunogenicity and Safety of Lyophilized Live-Attenuated Varicella Vaccine in Healthy Subjects Aged 13 to 55 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Shiyuan Wang, Department of epidemiology and biostatistics, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JSVCT058
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Chickenpox Vaccines
Keywords: clinical trial; phase 3; Immunogenicity; Safety; Live Attenuated Varicella Vaccine
MeSH Terms: interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Live Attenuated Varicella vaccine candidates (Experimental): freezedried live attenuated VarV developed by Beijing Minhai Biotechnology Co., LTD., which are derived from the Oka strain, cultured and harvested from inoculated MRC-5 human diploid cells inoculated human diploid cells (MRC-5), and then lyophilized with appropriate stabilizers.
  Interventions: Biological: Chickenpox Vaccines
- Marketed Live Attenuated Varicella vaccine (Active Comparator): the active control group received VarV produced by Changchun BCHT Biotechnology Co.,which are derived from human diploid cellsinoculated human diploid cells (MRC-5), and then lyophilized with appropriate stabilizers
  Interventions: Biological: Chickenpox Vaccines

INTERVENTIONS:
Biological: Chickenpox Vaccines — The vaccines require reconstitution with the provided sterile water for injection nd should be shaken well before use. Each human dose (0.5 ml) contains at least 3.3 log PFU of VZV.

SUMMARY:
Immunogenicity and Safety of a Live Attenuated Varicella Vaccine in Adolescents and adults Aged 13-55 Years: A Phase III, Randomized, Double-Blind, Active-Controlled Study

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged between 13 to 55 years who are permanent residents; Have obtained informed consent from the volunteer and/or their legal guardian, and signed the informed consent form; The volunteer and/or their legal guardian can comply with the requirements of the clinical trial protocol; Axillary temperature ≤37.0°C.

Exclusion Criteria:

* Females aged 18 to 55 years with a positive urine pregnancy test, pregnant women, women who are breastfeeding, or women planning to become pregnant within the next 3 months; Have a history of varicella vaccination, a history of chickenpox, or a history of herpes zoster infection; Allergic to known components of the study vaccine, or a history of severe allergic reactions to any vaccination; A history of epilepsy, seizures, or convulsions, or a family history of psychiatric disorders; Individuals with immunodeficiency, undergoing immunosuppressive therapy (e.g., oral corticosteroids), or having HIV-related immunocompromised status, or having close family members with congenital immune diseases; Have congenital malformations, developmental disorders, or severe chronic diseases (such as Down syndrome, diabetes, sickle cell anemia, neurological disorders, Guillain-Barré syndrome); Known or suspected concurrent diseases including: respiratory diseases, acute infections, or active chronic diseases, cardiovascular diseases, skin diseases, severe hypertension, or during treatment for malignant tumors; Diagnosed with coagulation dysfunction (such as coagulation factor deficiencies, coagulopathies, platelet abnormalities) or significant bruising or coagulation disorders; Have received blood products in the past 3 months; Have received live attenuated vaccines in the past 14 days or subunit or inactivated vaccines in the past 7 days; Have had various acute diseases or acute exacerbations of chronic diseases in the past 7 days; Have had a fever (axillary temperature ≥38.0°C) in the past 3 days; Any other factors deemed by the investigator as unsuitable for participation in the clinical trial.

Ages: 13 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1200 (Actual)
Dates: Start 2019-07-21 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-11-08 (Actual)

PRIMARY OUTCOMES:
seroconversion rate | 42 days after completing the full course of vaccination
  The primary immunogenicity endpoint was the seroconversion rate of VZV antibodies

SECONDARY OUTCOMES:
geometric mean titer (GMT) | 42 days after completing the full course of vaccination
  geometric mean titer (GMT) of VZV antibodies 42 days after vaccination
geometric mean fold increase (GMFI) | 42 days after completing the full course of vaccination
  geometric mean fold increase (GMFI) of VZV antibodies 42 days after vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Huaiyin District Center for Disease Control and prevention, Huaian, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Y, Wang S, Li G, Shi J, Chang X, Zhang H, Zhu F, Li J, Pan H, Sun J. Immunogenicity and safety of a live attenuated varicella vaccine in healthy subjects aged between 13 to 55 years: a double-blind, randomized, active-controlled phase III clinical trial in China. Expert Rev Vaccines. 2025 Dec;24(1):157-164. doi: 10.1080/14760584.2025.2457463. Epub 2025 Feb 7. PMID 39916494